CLINICAL TRIAL: NCT05440370
Title: Clinical Trial to Evaluate the Efficacy and Safety of MegaCarti® ; Cartilage Defect Treatment Assisting Cartilage Regeneration in Knee Cartilage Defects : Multicenter, Independent Evaluator and Subject Blinded, Microfracture Comparative, Superiority, Randomized, Confirmatory Clinical Study and 5 Years Follow up Study
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of MegaCarti® in Knee Cartilage Defects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: L&C Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LNC-MECA-001
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Cartilage Defects; microfracture; MegaCarti; cartilage regeneration
MeSH Terms: conditions — Osteoarthritis, Knee; Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MegaCarti® application after microfracture (Experimental): The experimental group is applied with MegaCarti® after microfracture. Afterwards, they visit at 6 weeks, 12 weeks, 24 weeks, and 48 weeks to conduct examinations and assess Questionnaires. Long-term follow-up Study is performed to subject that completes 48-week visit, at every 6 months for 5 years.
  Interventions: Device: MegaCarti®; Procedure: Microfracture
- Microfracture only (Active Comparator): The control group undergoes microfracture and they visit at 6 weeks, 12 weeks, 24 weeks, and 48 weeks after surgery to conduct examinations and assess Questionnaires.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Device: MegaCarti® — MegaCarti® application after microfracture through athroscopic or incision surgery
  Arms: MegaCarti® application after microfracture
Procedure: Microfracture — Microfracture through athroscopic or incision surgery

SUMMARY:
The MegaCarti® is the decellularized allogeneic cartilage and acts as a cover after bone marrow stimulation to prevent the loss of blood clots and induces cartilage regeneration by assisting in the location of stem cells derived from bone marrow.

The MegaCarti® is applied after Microfracture treatment on patients with Knee Cartilage Defects. The cartilage regeneration, which is a primary endpoint, is compared to the Microfracture group through MOCART evaluation. In addition, the improvement of pain and the recovery of Normal Range of motion are compared to the Microfracture group through secondary endpoints. Then, long-term follow-up study for 5 years is conducted to the experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years to 65 years
2. Patients or legal representatives who voluntarily decide to participate in the clinical trial, after which sign the consent form.
3. Defect: International Cartilage Repair Society(ICRS) Grade III or IV single defect chondral lesion on knee cartilage
4. Patients whose primary lesion site can be designated as one section of the knee joint, and the area can be determined as the main cause of clinical symptoms
5. knee cartilage defect size : Below 10 ㎠

Exclusion Criteria:

1. Patients who have autoimmune diseases (Ex. Rheumatoid arthritis)
2. Patients who underwent surgery related to cartilage defect treatment, such as microfracture, autologous chondrocyte therapy within the past 1 year (Possible for HTO surgery)
3. When screening, Patients who received intra-articular hyaluronic acid or steroid injections in the knee within 3 months
4. When screening, Patients who took oral steroid within 1 month
5. When screening, Patients who have clinically significant abnormalities in blood, serum, or urine tests
6. Patients taking immunosuppressive drug, or having immune disorder
7. Patients who can't take MRI scan
8. Patients with a history of cancer within the past five years
9. Patients who have chronic renal failure, active hepatitis, or poor blood sugar control
10. BMI index : 30 ㎏/㎡ or over
11. Patients who have gout or gout history in the knee
12. When screening, Women who are pregnant or breast-feeding, or women who are planning for pregnancy during the clinical trial, or women who have a possibility of pregnancy but do not use medically accepted methods of contraception.
13. Drug and alcohol addiction / dependence or mental disorder
14. Patients with risk factor for bleeding (Patients taking antithrombotic drugs other than aspirin)
15. Patients who have systemic or localized knee infection
16. Other than above, patients who are judged by medical investigator to be considered unsuitable for this clinical trial
17. Patients who participated in other clinical trials within three months before screening

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
MOCART score | 48 weeks after surgery
  Primary Endpoint [experimental group / control group]

SECONDARY OUTCOMES:
Comparison of IKDC score | Baseline and 12, 24, 48 weeks after surgery
  Secondary Endpoint [experimental group / control group]
Comparison of VAS score | Baseline and 6, 12, 24, 48 weeks after surgery
  Secondary Endpoint [experimental group / control group]
Comparison of KOOS score | Baseline and 12, 24, 48 weeks after surgery
  Secondary Endpoint [experimental group / control group]
Comparison of WOMAC score | Baseline and 12, 24, 48 weeks after surgery
  Secondary Endpoint [experimental group / control group]
Comparison of Kellgren-Lawrence grade | Baseline and 12, 24, 48 weeks after surgery
  Secondary Endpoint [experimental group / control group]
Frequency of rescue medication | For 48 weeks after surgery
  Secondary Endpoint [experimental group / control group]

CONTACTS AND LOCATIONS:
Overall Officials: Seong Hwan Kim, Professor, Principal Investigator — Yonsei University Health System, Gangnam Severance Hospital
Locations (4):
- South Korea (4):
  - National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Yonsei University Health System, Gangnam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No